CLINICAL TRIAL: NCT05351541
Title: A Double-blind, Randomized Trial Examining the Preliminary Efficacy of Psilocybin Therapy for People With Chronic Low Back Pain
Brief Title: Psilocybin Therapy for Chronic Low Back Pain
Acronym: POP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joshua Woolley, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Joshua Woolley, MD, PhD, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-21441
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic pain; Psilocybin; Psilocybin Therapy
MeSH Terms: conditions — Chronic Pain | interventions — Zolpidem; Modafinil

STUDY DESIGN:
Intervention Model Description: All patients will receive a dose of psilocybin between 1-30 mg, and one of the following: placebo, zolpidem, modafinial, or zolpidem and modafinil. All patients will receive two psilocybin preparation sessions , a single dose of psilocybin within a therapeutic environment (6-8 hours), three integration sessions and two follow up visits. All drugs will be orally administered during the dosing session. The study procedures will follow best practices for administering psilocybin in clinical trials.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial is testing various doses of psilocybin in combination with add-on medications. Participants, study staff and clinical assessors will be blinded to individual treatment conditions until study close-out. The clinician administered instruments will be administered by different clinical study staff than the facilitators who provide the preparation, psilocybin therapy, and integration sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Psilocybin in combination with Zolpidem and Modafinil (Experimental): Single dose of Psilocybin (1mg-30mg) in combination with zolpidem and modafinil
  Interventions: Drug: Psilocybin therapy with Zolpidem and Modafinil
- Psilocybin in combination with Zolpidem (Experimental): Single dose of Psilocybin (1mg-30mg) in combination with zolpidem
  Interventions: Drug: Psilocybin therapy with Zolpidem
- Psilocybin in combination with Modafinil (Experimental): Single dose of Psilocybin (1mg-30mg) in combination with modafinil
  Interventions: Drug: Psilocybin therapy with Modafinil
- Psilocybin in combination with Placebo (Experimental): Single dose of Psilocybin (1mg-30mg) in combination with placebo
  Interventions: Drug: Psilocybin therapy with Placebo

INTERVENTIONS:
Drug: Psilocybin therapy with Zolpidem and Modafinil — 1-30 mg (oral administration), Modafinil (oral administration), and Zolpidem (oral administration)
  Other Names: 4-phosphoryloxy- N,N-dimethyltryptamine
  Arms: Psilocybin in combination with Zolpidem and Modafinil
Drug: Psilocybin therapy with Zolpidem — 1-30 mg (oral administration), Zolpidem (oral administration), and placebo (oral administration)
  Other Names: 4-phosphoryloxy- N,N-dimethyltryptamine
  Arms: Psilocybin in combination with Zolpidem
Drug: Psilocybin therapy with Modafinil — 1-30 mg (oral administration), Modafinil (oral administration), and placebo (oral administration)
  Other Names: 4-phosphoryloxy- N,N-dimethyltryptamine
  Arms: Psilocybin in combination with Modafinil
Drug: Psilocybin therapy with Placebo — 1-30 mg (oral administration), and placebo (oral administration)
  Other Names: 4-phosphoryloxy- N,N-dimethyltryptamine
  Arms: Psilocybin in combination with Placebo

SUMMARY:
This study evaluates whether psilocybin therapy helps patients cope with chronic low back pain more effectively. Patients may be recruited at Stanford and University of California San Francisco (UCSF), study procedures will occur at UCSF. Each participant will receive a dose of psilocybin with possibly one or more other drugs. Participants will undergo two preparation sessions, a dosing session, three integration sessions to discuss their psilocybin experience, and several follow up sessions.

DETAILED DESCRIPTION:
Chronic pain is associated with higher levels of pain-related distress, depression, emotional dysfunction, helplessness, hopelessness, and suicidality. Psilocybin is a psychoactive drug that may be well-suited to easing the psychological and emotional symptoms of distress associated with chronic pain. Previous studies testing psilocybin therapy have shown improvements on multiple behavioral and psychiatric outcomes, but it is unknown whether psilocybin therapy similarly enables patients to cope with chronic pain more effectively. The investigators will determine whether psilocybin therapy improves patients' ability to cope with chronic low back pain. If psilocybin therapy is an effective treatment in this population, its use could be incorporated into interventions for chronic low back pain and other psychological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 70 years old
* Comfortable speaking and writing in English
* Diagnosed with chronic low back pain
* Able to attend all in-person visits at UCSF as well as virtual visits
* Has tried at least two previous medications/ procedures and physical therapy trials for low back pain

Exclusion Criteria:

* Chronic low back pain that is attributed to malignancy, subacute or acute fracture or infection
* Low back pain with radiation below the knee
* Low back pain with neurologic signs present
* Regular use of medications that may have problematic interactions with psilocybin, including but not limited to dopamine agonists, MAO inhibitors, antipsychotics, and stimulants
* A health condition that makes study unsafe or unfeasible, determined by study physicians

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in pain interference | Baseline, 1-month after psilocybin session
  The Brief Pain Inventory-Interference subscale (BPI) will be used to assess how pain interferes with a variety of daily activities (e.g., walking, lifting, mood, sleep, relationships). Seven items are rated on a scale from 0 (does not interfere) to 10 (completely interferes) for a total possible score ranging from 0 to 70. Higher scores represent greater interference from pain.

SECONDARY OUTCOMES:
Change in pain interference | Baseline, 1-week, and 3-months
  The Brief Pain Inventory-Interference subscale (BPI) will be used to assess how pain interferes with a variety of daily activities (e.g., walking, lifting, mood, sleep, relationships). Seven items are rated on a scale from 0 (does not interfere) to 10 (completely interferes) for a total possible score ranging from 0 to 70. Higher scores represent greater interference from pain.
Change in average pain intensity | Baseline, 1-week, 1-month, and 3-months after psilocybin session
  The Brief Pain Inventory with the Michigan Body Map will be used to assess pain location and worst, least, average, and present pain on a numerical rating scale from 0 (no pain) to 10 (pain as bad as you can imagine) over the past 24 hours, where higher scores represent greater pain intensity.
Change in clinical depressive symptom severity | Baseline, 1-week, 1-month, and 3-months after psilocybin session
  The 17-item clinician administered Hamilton Rating Scale for Depression will be used to assess changes in the severity of depressive symptoms. Each item is scored by a clinician on a 3- or 5-point scale from 0 (Not present) to 4 (severe) and summed for a total score between 0 and 52. A higher total score represents greater depressive symptom severity.
Change in depressive symptom severity | Baseline, pre-dosing session, 5-days, 11-days, and 77-days after psilocybin session
  The 7-item PROMIS-Depression self-report scale will be used as an additional indicator for changes in depression symptom severity. Items are endorsed on a 5-point scale ranging from 1 (Never) to 5 (Always). A higher total score represents greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Woolley, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided